CLINICAL TRIAL: NCT02011932
Title: Observational Study of Disease Progression and Risk Factors in Chronic Hepatitis C Caused by Plasma Donation
Brief Title: Prospective Observational Study of Disease Progression in Chronic Hepatitis C
Status: Active, not recruiting | Type: Observational
Sponsor: Beijing YouAn Hospital (Other)
Responsible Party: Principal Investigator, Zhongping Duan, Associate Dean,Professor,Chief Physician, Beijing YouAn Hospital
Other Study IDs: BJYAH-2011-045
Record Dates: First submitted 2013-12-06; First posted 2013-12-16 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Hepatitis C, Chronic; Disease Progression; Liver Cirrhosis
MeSH Terms: conditions — Hepatitis C, Chronic; Disease Progression; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma,liver biopsies specimens,
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy volunteers
- Chronic hepatitis C

SUMMARY:
The purpose of this study is to determine the progression of chronic hepatitis C patients infected by paid plasma donation,and explore the possible pathogenic mechanisms of disease progression in chronic hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* All these patients had a definite history of regular plasma donations with repeated blood cell re-transfusions.
* The Hepatitis C Virus antibody was positive.
* All patients did not receive interferon therapy before being recruited.

Exclusion Criteria:

* Patients with evidences for other forms of liver diseases.
* The coinfection with hepatitis B virus or other virus.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The plasma donors were primarily chosen from healthy farmers and agricultural workers living in a remote small city in the Northwest China.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2010-07; Primary Completion 2011-06 (Actual); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Fibrosis progression rate | 20 years
The incidence of cirrhosis | 20 years
Risk factors for the occurrence of cirrhosis | 20 years

SECONDARY OUTCOMES:
The incidence of hepatocellular carcinoma | 20 years
Number of participants with chronic hepatitis C-related complications | 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhongping Duan, Ph.D.,M.D., Principal Investigator — Beijing YouAn Hospital

REFERENCES:
- [Background] Seeff LB. Natural history of chronic hepatitis C. Hepatology. 2002 Nov;36(5 Suppl 1):S35-46. doi: 10.1053/jhep.2002.36806. PMID 12407575
- [Background] Poynard T, Bedossa P, Opolon P. Natural history of liver fibrosis progression in patients with chronic hepatitis C. The OBSVIRC, METAVIR, CLINIVIR, and DOSVIRC groups. Lancet. 1997 Mar 22;349(9055):825-32. doi: 10.1016/s0140-6736(96)07642-8. PMID 9121257
- [Background] Ghany MG, Kleiner DE, Alter H, Doo E, Khokar F, Promrat K, Herion D, Park Y, Liang TJ, Hoofnagle JH. Progression of fibrosis in chronic hepatitis C. Gastroenterology. 2003 Jan;124(1):97-104. doi: 10.1053/gast.2003.50018. PMID 12512034
- [Background] Seeff LB, Miller RN, Rabkin CS, Buskell-Bales Z, Straley-Eason KD, Smoak BL, Johnson LD, Lee SR, Kaplan EL. 45-year follow-up of hepatitis C virus infection in healthy young adults. Ann Intern Med. 2000 Jan 18;132(2):105-11. doi: 10.7326/0003-4819-132-2-200001180-00003. PMID 10644270